CLINICAL TRIAL: NCT02777138
Title: Impact of Ageing on Adipose, Muscle and Systemic Inflammation
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Bath (Other)
Responsible Party: Principal Investigator, William Trim, Ph.D. Student, University of Bath
Other Study IDs: 16/sw/0003
Record Dates: First submitted 2016-05-06; First posted 2016-05-19 (Estimated); Last update posted 2018-08-24 (Actual); Status verified 2018-08

CONDITIONS: Inflammation; Aging
Keywords: Adipose tissue; Inflammation; Age Comparison; Macrophages; T-lymphocytes; Adipose Progenitors
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — muscle and adipose biopsies blood plasma blood serum peripheral blood mononuclear cells
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Young males aged 20-35 years old: Maintaining a normal daily living lifestyle
  * Healthy
  * Reasonably active- PAL: 1.4-1.9
  * Non-obese- Fat mass index based on DEXA of 4-8kg/m2
  * Weight stable for more than 3 months (±3% body mass)
  * Non-smoker
  * No chronic illness, cardiac, pulmonary, liver, or kidney abnormalities, uncontrolled hypertension, peripheral arterial disease, insulin- or non-insulin dependent diabetes or other metabolic disorders
  * No daily consumption of analgesic or anti-inflammatory drug(s) including NSAIDs and corticosteroids, prescription or non-prescription
  * No medications that may influence lipid or carbohydrate metabolism or immune system function
  * No known negative reaction to lidocaine
  * No participation in heavy resistance training
  Interventions: Other: Maintaining a normal daily living lifestyle
- Old males aged 65-85 years old: Maintaining a normal daily living lifestyle
  * Healthy
  * Reasonably active- PAL: 1.4-1.9
  * Non-obese- Fat mass index based on DEXA of 4-8kg/m2
  * Weight stable for more than 3 months (±3% body mass)
  * Non-smoker
  * No chronic illness, cardiac, pulmonary, liver, or kidney abnormalities, uncontrolled hypertension, peripheral arterial disease, insulin- or non-insulin dependent diabetes or other metabolic disorders
  * No daily consumption of analgesic or anti-inflammatory drug(s) including NSAIDs and corticosteroids, prescription or non-prescription
  * No medications that may influence lipid or carbohydrate metabolism or immune system function
  * No known negative reaction to lidocaine
  * No participation in heavy resistance training
  Interventions: Other: Maintaining a normal daily living lifestyle

INTERVENTIONS:
Other: Maintaining a normal daily living lifestyle — participants will undertake a normal lifestyle with no alterations to daily living in order to access the differences in tissue (muscle and adipose) and systemic inflammation between the two age cohorts

SUMMARY:
The accumulation and dysfunction of excess adipose (fat) tissue that occurs with ageing is associated with a number of chronic inflammatory disorders such as type 2 diabetes and cardiovascular disease but the underlying mechanisms are not understood.

DETAILED DESCRIPTION:
Adipose tissue is a highly dynamic organ that produces a wide array of adipokines which can affect the function of other tissues throughout the body. The physiology of adipose tissue is a relatively new and exciting area of research and researchers are learning more about its complexity, in particular the way in which adipose tissue plays a dynamic and active role in various normal and pathological processes. Comparatively little is known about the changes that occur within adipose tissue over the natural course of ageing - and adipose dysfunction could play a role in ageing-related chronic systemic inflammatory diseases such as type 2 diabetes and cardiovascular disease.

In this study, the investigators would like to investigate inflammatory and metabolic changes that occur within adipose tissue with ageing. the investigators would also like to examine whether age-related changes in adipose tissue are specific to this particular tissue type by comparing adipose-resident immune cell populations and measures of inflammation and metabolism to those in muscle tissue and blood.

By exploring the immune dysfunction that occurs with ageing in adipose tissue and relating them to inflammatory and metabolic differences in muscle and blood, this work may potentially reveal causal mechanisms in the development of ageing-related chronic inflammatory diseases and ultimately lead to the development of better treatment/management strategies.

BACKGROUND Adipose tissue is sizeable endocrine organ and is highly dynamic, producing a wide array of adipokines which can affect a range of physiological processes including regulation of appetite, energy expenditure, insulin sensitivity, inflammation, endocrine and reproductive systems and bone metabolism. Ageing is a process that is associated with adipose tissue accumulation, changes in adipose tissue distribution and its dysfunction which in turn are linked to the development of chronic inflammatory disorders such as type 2 diabetes and cardiovascular disease.

Adipose tissue inflammation may be key Adipose tissue consists not only of adipocytes, but also many other cell types including endothelial cells, preadipocytes, immune cells such as macrophages and lymphocytes such that adipocytes themselves may only represent 60-70 % cell numbers in adipose tissue. Research from over the last decade or so suggests that the presence of immune cells within the adipose tissue itself are important in regulating both local and systemic inflammation/production of adipokines. For example, adipose tissue macrophages contribute the majority of the pro-inflammatory cytokine TNFα and ~50% IL6 secreted by adipose tissue, which show increased secretion with adipose tissue dysfunction and are implicated in the development of chronic inflammatory disorders. Changes in adipose resident immune cells have been relatively well studied in obesity but there are comparatively few studies in humans examining changes in immune cell populations and their potential impact on adipose tissue inflammation in the context of ageing. Given the time-course of adipose tissue accumulation in obesity compared to ageing, there is the potential for differences in the underlying mechanisms of adipose tissue dysfunction to occur.

In humans, there is overwhelming evidence (including work by the investigator's group) that macrophages accumulate in subcutaneous adipose tissue with obesity and are important mediators of adipose tissue inflammation. Additionally, work performed by this group has also shown that T cells in adipose tissue are more activated with obesity and this may also be related to levels of adipose tissue inflammation. Only one study has attempted to investigate the impact of ageing on immune cells in adipose tissue, however, this was in a very specific population (Pima Indians) and only up-to the age of 45 years so it is not known how immune cells change with further increases in age where chronic inflammatory disorders become more prevalent. Studies using mouse models indeed suggest that there are discrepancies in immune cell populations within adipose tissue following diet-induced obesity compared to ageing. In mice, it is not clear if there is a change in the number or just a change from an anti- to pro-inflammatory phenotype which would be in contrast to obesity, where there is evidence of both an increase in number and skewing towards a pro-inflammatory phenotype. Mice also show an increase in T-cells in adipose tissue with ageing - especially in T-regulatory cells, however, in diet-induced obesity there may be an increase in the number of pro-inflammatory effector cells (e.g. CD8+).

The potential role of adipose tissue inflammation in the development of age-related chronic inflammatory disorders and how this compares to the investigators' previous work in the context of obesity is something the investigators are keen to address in the present study.

Investigating tissue specific changes with ageing With ageing there is an increased deposition of adipose tissue within muscle and this can have profound effects on muscle tissue including inducing insulin resistance and lipotoxicity. Considering that muscle is one of the major sites for glucose uptake, impairment in this process can have a profound effect on systemic glucose concentrations and whole body insulin resistance. Like adipose tissue, muscle itself is host to resident immune cells, but it is not known whether these differ in terms of proportion or function to those found in adipose tissue. Furthermore, it is not known how these immune cells in muscle tissue may affect local and systemic inflammation in the development of ageing-related chronic inflammatory diseases. It is important to consider the role of different tissues in disorders that affect the body as a whole as there may be specific responses to ageing that need to be considered when trying to understand the underlying pathophysiology of ageing-related chronic diseases. Thus, the impact of ageing on muscle immune cells and inflammation is another factor that the investigators are keen to address in the present study. the investigators are especially interested in examining whether ageing affects adipose and muscle in a similar or different way.

Purpose The purpose of this study is to investigate inflammatory and metabolic changes in adipose tissue that occur with ageing and to compare these changes to those in muscle and blood.

By comparing metabolic and inflammatory parameters within adipose tissue, muscle and the circulation in younger and older individuals, the investigators hope to gain vital clues regarding the potential pathogenic mechanisms involved in the development of ageing-related chronic inflammatory diseases. With greater understanding of these mechanisms the investigators hope to prepare the ground for new and more effective means of prevention/treatments for ageing-related chronic inflammatory diseases.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Aged between 20-35 years (Group 1) or 65-85 years (Group 2)
* Fat mass index based on DEXA between 4-8 kg/m2
* Weight stable for more than 3 months (no change in weight +/- 3%)
* Physical Activity Level (PAL) between 1.4 and 1.9
* Non-smoker
* Healthy

Exclusion Criteria:

* Any chronic illness, cardiac, pulmonary, liver, or kidney abnormalities, uncontrolled hypertension, peripheral arterial disease, insulin- or non-insulin dependent diabetes or other metabolic disorders
* Individuals who consume on a daily basis any analgesic or anti-inflammatory drug(s) including NSAIDs and corticosteroids, prescription or non-prescription
* Taking any medications that may influence lipid or carbohydrate metabolism or immune system function
* Individuals with a known negative reaction to lidocaine anaesthetic
* Participation in heavy resistance training

Ages: 20 Years to 85 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: general free-living public in the Bath and the surrounding areas
Sampling Method: Non-Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2016-05; Primary Completion 2018-03 (Actual); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
Differences in immune cell populations (macrophages/Tcells) in adipose tissue of young versus old males | through to study completion, an average of 14 months

SECONDARY OUTCOMES:
the impact of ageing on mRNA expression of key metabolic and inflammatory genes in adipose tissue. | through to study completion, an average of 14 months
the impact of ageing on metabolic and inflammatory protein secretions (into culture media) from adipose tissue | through to study completion, an average of 14 months
differences in immune cell populations in muscle tissue and blood compared to adipose tissue from the same individuals and the impact of ageing on immune cell populations in muscle tissue. | through to study completion, an average of 14 months
the impact of ageing on mRNA expression of other key metabolic and inflammatory genes in muscle tissue. | through to study completion, an average of 14 months
activation/inhibition of e.g. insulin stimulated pathways in adipose and muscle tissues (for example assessment of Akt/IRS1 phosphorylation by western blot analysis). | through to study completion, an average of 14 months

CONTACTS AND LOCATIONS:
Overall Officials: Dylan Thompson, Professor, Principal Investigator — University of Bath
Locations (1):
- university of bath - Department for Health, Bath, Somerset, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Alderete TL, Sattler FR, Sheng X, Tucci J, Mittelman SD, Grant EG, Goran MI. A novel biopsy method to increase yield of subcutaneous abdominal adipose tissue. Int J Obes (Lond). 2015 Jan;39(1):183-6. doi: 10.1038/ijo.2014.90. Epub 2014 May 21. PMID 24849392
- [Background] Bourlier V, Zakaroff-Girard A, Miranville A, De Barros S, Maumus M, Sengenes C, Galitzky J, Lafontan M, Karpe F, Frayn KN, Bouloumie A. Remodeling phenotype of human subcutaneous adipose tissue macrophages. Circulation. 2008 Feb 12;117(6):806-15. doi: 10.1161/CIRCULATIONAHA.107.724096. Epub 2008 Jan 28. PMID 18227385
- [Background] Cancello R, Tordjman J, Poitou C, Guilhem G, Bouillot JL, Hugol D, Coussieu C, Basdevant A, Bar Hen A, Bedossa P, Guerre-Millo M, Clement K. Increased infiltration of macrophages in omental adipose tissue is associated with marked hepatic lesions in morbid human obesity. Diabetes. 2006 Jun;55(6):1554-61. doi: 10.2337/db06-0133. PMID 16731817
- [Background] Clement K, Viguerie N, Poitou C, Carette C, Pelloux V, Curat CA, Sicard A, Rome S, Benis A, Zucker JD, Vidal H, Laville M, Barsh GS, Basdevant A, Stich V, Cancello R, Langin D. Weight loss regulates inflammation-related genes in white adipose tissue of obese subjects. FASEB J. 2004 Nov;18(14):1657-69. doi: 10.1096/fj.04-2204com. PMID 15522911
- [Background] Curat CA, Miranville A, Sengenes C, Diehl M, Tonus C, Busse R, Bouloumie A. From blood monocytes to adipose tissue-resident macrophages: induction of diapedesis by human mature adipocytes. Diabetes. 2004 May;53(5):1285-92. doi: 10.2337/diabetes.53.5.1285. PMID 15111498
- [Background] Dyck DJ, Heigenhauser GJ, Bruce CR. The role of adipokines as regulators of skeletal muscle fatty acid metabolism and insulin sensitivity. Acta Physiol (Oxf). 2006 Jan;186(1):5-16. doi: 10.1111/j.1748-1716.2005.01502.x. PMID 16497175
- [Background] Fabbrini E, Cella M, McCartney SA, Fuchs A, Abumrad NA, Pietka TA, Chen Z, Finck BN, Han DH, Magkos F, Conte C, Bradley D, Fraterrigo G, Eagon JC, Patterson BW, Colonna M, Klein S. Association between specific adipose tissue CD4+ T-cell populations and insulin resistance in obese individuals. Gastroenterology. 2013 Aug;145(2):366-74.e1-3. doi: 10.1053/j.gastro.2013.04.010. Epub 2013 Apr 15. PMID 23597726
- [Background] Fantuzzi G. Adipose tissue, adipokines, and inflammation. J Allergy Clin Immunol. 2005 May;115(5):911-9; quiz 920. doi: 10.1016/j.jaci.2005.02.023. PMID 15867843
- [Background] Goossens GH, Blaak EE, Theunissen R, Duijvestijn AM, Clement K, Tervaert JW, Thewissen MM. Expression of NLRP3 inflammasome and T cell population markers in adipose tissue are associated with insulin resistance and impaired glucose metabolism in humans. Mol Immunol. 2012 Mar;50(3):142-9. doi: 10.1016/j.molimm.2012.01.005. Epub 2012 Feb 8. PMID 22325453
- [Background] Lumeng CN, Liu J, Geletka L, Delaney C, Delproposto J, Desai A, Oatmen K, Martinez-Santibanez G, Julius A, Garg S, Yung RL. Aging is associated with an increase in T cells and inflammatory macrophages in visceral adipose tissue. J Immunol. 2011 Dec 15;187(12):6208-16. doi: 10.4049/jimmunol.1102188. Epub 2011 Nov 9. PMID 22075699
- [Background] Nishimura S, Manabe I, Nagasaki M, Eto K, Yamashita H, Ohsugi M, Otsu M, Hara K, Ueki K, Sugiura S, Yoshimura K, Kadowaki T, Nagai R. CD8+ effector T cells contribute to macrophage recruitment and adipose tissue inflammation in obesity. Nat Med. 2009 Aug;15(8):914-20. doi: 10.1038/nm.1964. Epub 2009 Jul 26. PMID 19633658
- [Background] Ortega Martinez de Victoria E, Xu X, Koska J, Francisco AM, Scalise M, Ferrante AW Jr, Krakoff J. Macrophage content in subcutaneous adipose tissue: associations with adiposity, age, inflammatory markers, and whole-body insulin action in healthy Pima Indians. Diabetes. 2009 Feb;58(2):385-93. doi: 10.2337/db08-0536. Epub 2008 Nov 13. PMID 19008342
- [Background] Pararasa C, Bailey CJ, Griffiths HR. Ageing, adipose tissue, fatty acids and inflammation. Biogerontology. 2015 Apr;16(2):235-48. doi: 10.1007/s10522-014-9536-x. Epub 2014 Nov 4. PMID 25367746
- [Background] Thompson D, Karpe F, Lafontan M, Frayn K. Physical activity and exercise in the regulation of human adipose tissue physiology. Physiol Rev. 2012 Jan;92(1):157-91. doi: 10.1152/physrev.00012.2011. PMID 22298655
- [Background] Travers RL, Motta AC, Betts JA, Bouloumie A, Thompson D. The impact of adiposity on adipose tissue-resident lymphocyte activation in humans. Int J Obes (Lond). 2015 May;39(5):762-9. doi: 10.1038/ijo.2014.195. Epub 2014 Nov 12. PMID 25388403
- [Background] Trayhurn P, Drevon CA, Eckel J. Secreted proteins from adipose tissue and skeletal muscle - adipokines, myokines and adipose/muscle cross-talk. Arch Physiol Biochem. 2011 May;117(2):47-56. doi: 10.3109/13813455.2010.535835. Epub 2010 Dec 15. PMID 21158485
- [Background] Varma V, Yao-Borengasser A, Rasouli N, Nolen GT, Phanavanh B, Starks T, Gurley C, Simpson P, McGehee RE Jr, Kern PA, Peterson CA. Muscle inflammatory response and insulin resistance: synergistic interaction between macrophages and fatty acids leads to impaired insulin action. Am J Physiol Endocrinol Metab. 2009 Jun;296(6):E1300-10. doi: 10.1152/ajpendo.90885.2008. Epub 2009 Mar 31. PMID 19336660
- [Background] Weisberg SP, McCann D, Desai M, Rosenbaum M, Leibel RL, Ferrante AW Jr. Obesity is associated with macrophage accumulation in adipose tissue. J Clin Invest. 2003 Dec;112(12):1796-808. doi: 10.1172/JCI19246. PMID 14679176
- [Background] Zeyda M, Farmer D, Todoric J, Aszmann O, Speiser M, Gyori G, Zlabinger GJ, Stulnig TM. Human adipose tissue macrophages are of an anti-inflammatory phenotype but capable of excessive pro-inflammatory mediator production. Int J Obes (Lond). 2007 Sep;31(9):1420-8. doi: 10.1038/sj.ijo.0803632. Epub 2007 Jun 26. PMID 17593905
- [Background] Xu H, Barnes GT, Yang Q, Tan G, Yang D, Chou CJ, Sole J, Nichols A, Ross JS, Tartaglia LA, Chen H. Chronic inflammation in fat plays a crucial role in the development of obesity-related insulin resistance. J Clin Invest. 2003 Dec;112(12):1821-30. doi: 10.1172/JCI19451. PMID 14679177